CLINICAL TRIAL: NCT03437252
Title: The Association of Physical Activity With Readmission Due to Exacerbation in COPD Patients
Brief Title: Physical Activity in Chronic Obstructive Pulmonary Disease(COPD) Acute Exacerbation Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hye Yun Park, Associate Professor, Samsung Medical Center
Other Study IDs: 2017-11-009-002
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: COPD Exacerbation
Keywords: Chronic obstructive pulmonary disease; Chronic obstructive pulmonary disease acute exacerbation; Physical activity; Wearable arm device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who are suffering from Chronic Obstructive Pulmonary Disease (COPD) had a decreased level of physical activity which is consequentially related to another acute exacerbation event. In this study, we selected patients from those who were admitted for acute exacerbation of COPD, evaluated physical activity by accelerometer (wearable multisensory armband devices) to find out the correlation between physical activity in COPD acute exacerbation patients.

ELIGIBILITY:
Inclusion Criteria:

* COPD patient who have forced expiratory volume in one second/ forced vital capacity (FEV1/FVC) < 70% by spirometry and those who have not been admitted for acute exacerbation in recent 3 months

Exclusion Criteria:

* Those who does not consent or those who have drug addiction, psycho-socially or medically not feasible to this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on COPD patients who visited Samsung medical center.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2025-11-19 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Re admission rate after COPD acute exacerbation | 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea